CLINICAL TRIAL: NCT03556826
Title: Feasibility and Preliminary Efficacy of Social Value Training in Toddlers With Elevated Autism Symptoms
Brief Title: Social Value Training in Toddlers With Elevated Autism Symptoms
Acronym: SVT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was hindered by Covid and masking, therefore was unable to be completed as intended.
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000021541; P50MH115716 (NIH); 1R01MH124892-01A1 (NIH)
Record Dates: First submitted 2018-06-01; First posted 2018-06-14 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social Value Learning (Experimental): For each child, two faces, randomly selected from the pool of four faces, will be assigned the high-value (HV) status and the other two the low-value (LV) status. Value status will be randomized between the faces and children and all four faces will have the same probability of being assigned HV or LV across all participants. A gaze fixation on a HV face will always activate a dynamic display and the face will smile brightly. A gaze fixation on a LV face will always result in no change to its display. Effects of training will be tested one day (efficacy) and one month (maintenance) after training. During each of the follow-up assessments, each child will first undergo the Laboratory Selective Attention (LSA) task to assess if they retained value-face associations from the training sessions, followed by the Real-World Selective Attention (RWSA) task to evaluate generalization.
  Interventions: Behavioral: Social Value Learning Training

INTERVENTIONS:
Behavioral: Social Value Learning Training — For each child, two faces will be assigned the high-value (HV) status and the other two the low-value (LV) status. Value status will be randomized between the faces and children and all four faces will have the same probability of being assigned HV or LV across all participants. A gaze fixation on a HV face will always activate a dynamic display and the face will smile brightly. A gaze fixation on a LV face will always result in no change to its display.

SUMMARY:
In the proposed pilot study, ASD+ toddlers will undergo Social Value Training (SVT) using a gaze-contingent eye-tracking paradigm in toddlers with elevated symptoms of ASD (ASD+) (n=48). SVT will be administered over a two-day period and the training effects will be assessed by changes in visual attention to high-value (HV) faces as compared to low-value (LV) faces between baseline, post-baseline, and a follow-up assessment using two tasks: a laboratory selective attention (LSA) task and real-world selective attention (RWSA) task. The investigators will also evaluate acceptability and feasibility of the value training and contribution of sex, nonverbal developmental level, and severity of autism symptoms to response to the training.

DETAILED DESCRIPTION:
One of the markers of autism spectrum disorders (ASD) in infants and toddlers is impaired selective attention to faces. This impairment diminishes their ability to learn from and interact adaptively with others in real-world environments. Attentional selection in the social domain relies, in part, on one's ability to encode reward values of people and store these values in long-term memory as stable values. The 'stable' values (henceforth, 'values') are learned over the course of repeated learning opportunities, and once acquired, they are signaled rapidly, preferentially directing gaze to encoded faces of importance (high-value, HV) based on their hedonic or informative properties in the past. Automatic responses based on values stored in long-term memory are essential for survival when decisions have to be made rapidly (e.g., mother versus stranger). Learning about values is subserved by the reward learning system in the brain involving basal ganglia (BG) circuitry. This circuitry is implicated in the pathophysiology of ASD and extant evidence suggests that individuals with ASD exhibit specific impairments in learning the reward value of social stimuli such as faces. Based on this evidence, the investigators propose that limited attention to faces in toddlers with elevated autism symptoms (ASD+) is, in part, driven by impaired value learning in the social domain, affecting their ability to rapidly and preferentially select HV faces and ignore low-value (LV) faces in the complex real-world environment. Consequently, they exhibit diminished spontaneous attention to faces in general, and when they look at faces, they may distribute their limited attentional resources between high- (e.g., mother or therapist) and low-value (stranger) individuals in a trial-and-error fashion. The investigators further hypothesize that reinforcing attention of children with ASD+ toward specific faces through social value training (SVT) will increase their attention to these faces in real-world environments. In the proposed pilot study, ASD+ toddlers will undergo Social Value Training (SVT) using a gaze-contingent eye-tracking paradigm in toddlers with elevated symptoms of ASD (ASD+) (n=48). SVT will be administered over a two-day period and the training effects will be assessed by changes in visual attention to high-value (HV) faces as compared to low-value (LV) faces between baseline, post-baseline, and a follow-up assessment using two tasks: a laboratory selective attention (LSA) task and real-world selective attention (RWSA) task. The investigators will also evaluate acceptability and feasibility of the value training and contribution of sex, nonverbal developmental level, and severity of autism symptoms to response to the training.

Study was hindered by Covid and masking, therefore primary and secondary outcomes were unable to be collected as intended.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age of 37-42 weeks
* Appropriate weight for gestational age
* Presence of an older full biological sibling with ASD
* Autism Diagnostic Observation Schedule-2 (ADOS-2) score at 18 months in the clinical range (calibrated severity score >3)

Exclusion Criteria:

* Congenital infections
* Non-febrile seizure disorder
* Hearing loss
* Visual impairment
* Presence of any known chromosomal abnormality or congenital infection
* Prenatal exposure to illicit drugs
* Major psychotic disorder in first degree relatives.

Ages: 15 Months to 21 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Proportion of looking at faces during the laboratory and real-world tests | Average trial duration: for laboratory task: 2 seconds, for real-world task: 1 minute
  The proportion of time spent attending to faces assigned HV and LV, standardized by the amount of valid eye-tracking data collected during the trial

SECONDARY OUTCOMES:
Proportion of looking at the scene during laboratory and real-world tests | Average trial duration: for laboratory task: 2 seconds, for real-world task: 1 minute
  The proportion of valid eye tracking time collected during test trials standardized over the test trials duration

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Chawarska, PhD, Principal Investigator — Social and Affective Neuroscience of Autism Program, Yale Child Study Center
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No